CLINICAL TRIAL: NCT02429466
Title: Phase I Study of the Hypomethylating Drug SGI-110 Plus Cisplatin in Relapsed Refractory Germ Cell Tumors
Brief Title: Study of the Hypomethylating Drug Guadecitabine (SGI-110) Plus Cisplatin in Relapsed Refractory Germ Cell Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nasser Hanna (Other)
Responsible Party: Sponsor-Investigator, Nasser Hanna, Assistant Professor of Clinical Medicine, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUCRO-0508; 1502729080 (Other: Indiana University IRB)
Record Dates: First submitted 2015-04-14; First posted 2015-04-29 (Estimated); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Germ Cell Tumor; Testis Cancer; Testicular Cancer
Keywords: testicular germ cell tumor; ovarian germ cell tumor; platinum refractory; cisplatin; SGI110; Guadecitabine
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal; Testicular Neoplasms; Testicular Germ Cell Tumor | interventions — guadecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Guadecitabine (SGI-110) (Experimental)
  Interventions: Drug: Guadecitabine (SGI-110)

INTERVENTIONS:
Drug: Guadecitabine (SGI-110) — SGI-110 will be given subcutaneously, daily, 30 mg/m2 on days (1-5) followed by cisplatin 100mg/m2 on day 8 every 4 weeks.
  Other Names: Guadecitabine

SUMMARY:
This is an open-label, single arm, Phase I dose escalation study in subjects with refractory germ cell tumor (rGCT). This phase I will evaluate the safety and efficacy of SGI-110 in combination with cisplatin in subjects with rGCT. The primary objective is to determine the maximum tolerated dose (MTD) of SGI-110 to be used prior to cisplatin. A total of 15 subjects will be enrolled in this study at the Indiana University Simon Cancer Center.

DETAILED DESCRIPTION:
Primary Objective:

To assess the safety and toxicity of guadecitabine (SGI-110) plus cisplatin including the dose limiting toxicity (DLT) and to determine the Maximum tolerated dose (MTD)

Secondary Objective:

To assess the efficacy of guadecitabine (SGI-110) to resume sensitivity to cisplatin in refractory GCT

Correlative Objective:

To evaluate the pharmacodynamic activity of guadecitabine (SGI-110) Evaluate miRNA biomarkers in serum on day 1 of cycles 1-6

Intervention and Mode of Delivery: Guadecitabine (SGI-110) will be given subcutaneously, daily, 30 mg/m2 on days (1-5) followed by cisplatin 100mg/m2 on day 8 every 4 weeks.

Duration of Intervention and Evaluation:

Treatment will be continued for a maximum of 6 cycles or until disease progression or unacceptable toxicity whichever occurs first. Subjects who are responding to therapy without major toxicty would be allowed to continue on single agent guadecitabine (SGI-110) at the MTD after 4-6 cycles of the combination therapy until disease progression. Subjects will be followed after the last cycle every 2 months for the 1st year, and every 4 months thereafter until death (expected overall survival less than 12 months).

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old at the time of informed consent
2. Written informed consent and HIPAA authorization for release of personal health information.
3. Subjects who are willing and able to comply with the protocol and study procedures including willingness to undergo tumor biopsy for tumor cells before therapy at Cycle 1, Day 1, and Day 8 (before cisplatin dose) if this is clinically and safely feasible to do so.
4. Subjects with histologically or serologically confirmed diagnosis of recurrent germ cell tumor.
5. Subjects who have platinum-resistant disease. There is no limit on the number of prior treatment regimens.
6. Subjects must have had prior high dose chemotherapy (HDCT) treatment when indicated.
7. Subjects who have measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or elevated Tumor markers (hCG or AFP).

   Note: patients without measurable disease are allowed on the study as long as they have clearly rising tumor markers and they will be exempt from biopsy.
8. Subjects with ECOG performance status of 0-2.
9. Subjects must be at least 3 weeks from last chemotherapy.
10. Females of childbearing potential must not be pregnant or breast-feeding. Male and female patients of reproductive potential must agree to use two forms of highly effective contraception from the screening visit through 30 days after the last dose of study drug. Acceptable forms of effective contraception include:

    * Oral, injected or implanted hormonal methods of contraception.
    * Placement of an intrauterine device (IUD) or intrauterine system (IUS).
    * Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.
    * Male sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate).
    * True abstinence: When this is in line with the preferred and usual lifestyle of the subject. [Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.] Pregnancy tests for females of childbearing potential are required; must be serum at screening and the post treatment safety assessment visit. A positive urine pregnancy test must be confirmed by a serum pregnancy test and a pelvic US since some NSGCT may secrete beta-hCG and cause a false positive pregnancy. A pelvic US does not need to be repeated with each cycle unless the treating physician thinks it is necessary to do so.
11. The following laboratory values must be obtained within 14 days prior to registration for protocol therapy.

    * Absolute neutrophil count ≥ 1500 cells/mm3
    * Hemoglobin (Hgb) ≥ 8 g/dL
    * Platelets count ≥ 100,000 cells/mm3
    * Serum creatinine levels ≤ 1.5 mg/dl and calculated (by Cockcroft-Gault formula) or measured creatinine clearance ≥ 50 mL/min
    * Bilirubin ≤ 2 x ULN
    * Aspartate aminotransferase (AST, SGOT) ≤ 3 x ULN
    * Alanine aminotransferase (ALT, SGPT) ≤ 3 x ULN

Exclusion Criteria:

1. Active central nervous system (CNS) metastases. Subjects with neurological symptoms should undergo a head CT scan or brain MRI to exclude brain metastasis, at the discretion of the treating physician.

   NOTE: A subject with prior brain metastasis may be considered if they have completed their treatment for brain metastasis, no longer require corticosteroids, and are asymptomatic.
2. Treatment with any investigational agent within 30 days prior to registration for protocol therapy.
3. Concurrent participation in a clinical trial which involves another investigational agent.
4. Subjects with Grade 2 or greater neuropathy.
5. Subjects with a life-threatening illness, medical condition or organ system dysfunction, or other reasons which, in the Investigator's opinion, could compromise the subject's safety, interfere with or compromise the integrity of the study outcomes including incomplete recovery from the acute effects from any prior anti-neoplastic therapy.
6. Pregnancy or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-04-27 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2019-02-13 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) of guadecitabine (SGI-110) plus cisplatin | During chemotherapy (weeks 1-18)
Maximum tolerated dose (MTD) of SGI-110 plus cisplatin | During chemotherapy (weeks 1-18)

SECONDARY OUTCOMES:
Objective response rate (ORR) | Days 42, 84, 126, 159, and 220
  To evaluate Objective response rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST)
Progression free survival (PFS) | Days 42, 84, 126, 159, and 220
  The investigators will look at the duration between starting the therapy until progression of disease of subjects on this study

OTHER OUTCOMES:
Pharmacodynamic activity of SGI-110 | Day 8
  Blood collection to measure change in peripheral blood mononuclear cells (PBMCs), global DNA and selected genes, and expression of DNMT levels
Pharmacodynamic activity of SGI-110 | Day 8
  Tumor tissue collection to measure change in global DNA and selected tumor genes, and expression of DNMT levels

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Hanna, MD, Principal Investigator — Indiana University School of Medicine
Locations (2):
- United States (2):
  - Indiana University Hospital, Indianapolis, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana